CLINICAL TRIAL: NCT02252809
Title: An Open-Label, Parallel Group, Controlled Study in Healthy Subjects to Characterize Biological Responses to Immunological Challenges and to Measure the Effect of Marketed Anti-Inflammatory Agents on Those Responses
Brief Title: Effect of Anti-Inflammatory Agents on Biological Responses to Endotoxin Inhalation in Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Michel, Chief of Department, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FXT-01; FXT-01 (Other: CHU Brugmann)
Record Dates: First submitted 2014-09-23; First posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Innate Immunity
Keywords: inflammation endotoxin anti-TNF corticosteroids
MeSH Terms: interventions — Adalimumab; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- adalimumab (Active Comparator): adalimumab 40 mg by subcutaneous way 7 days before endotoxin inhalation
  Interventions: Drug: adalimumab
- methylprednisolone (Active Comparator): methylprednisolone 20 mg daily , 7 days before endotoxin inhalation
  Interventions: Drug: methylprednisolone
- control (No Intervention): no intervention, 7 days before endotoxin inhalation

INTERVENTIONS:
Drug: adalimumab
  Arms: adalimumab
Drug: methylprednisolone
  Arms: methylprednisolone

SUMMARY:
The main objective of this study is to characterize the biological responses elicited by endotoxin inhalation applied to healthy subjects, and to assess the effect of standard anti-inflammatory agents (i.e. adalimumab and methylprednisolone) on these biological responses.

DETAILED DESCRIPTION:
This open-label, single-center, parallel-group clinical trial is designed to evaluate Humira® or methylprednisolone versus no treatment in healthy subjects applied inhaled endotoxin challenges.

A total of 30 healthy adult subjects who meet all inclusion and exclusion criteria will be randomised in a 1:1:1 ratio to one of the following cohorts:

* Cohort 1 subjects receive no study drug during the study.
* Cohort 2 subjects receive an oral 7-day course of the corticosteroid (methylprednisolone) during the study, starting on study Day 1. The daily dose is 20 mg.
* Cohort 3 subjects receive a single subcutaneous injection of the anti-tumor necrosis factor (TNF) (adalimumab) on study Day 1, administered as a 40 mg dose.

The study will include a Screening period of up to 21 days, during which subject eligibility will be assessed and Screening responses to endotoxin exposure challenge will be collected. Eligible subjects will initially undergo an 8-day treatment period, during which they will receive treatment based on their assigned cohort (or will receive no treatment if assigned to Cohort 1) and will be applied with the endotoxin challenges. After the treatment period, subjects will be followed up until study Day 42.

Efficacy evaluations will include specific responses to endotoxin challenge, and effects of methylprednisolone and adalimumab on these responses. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 49 years, inclusive.
2. Responsive to inhaled endotoxin; defined as a reduction of 10% or greater in forced expiratory volume in 1 second (FEV1) following inhalation of 20 µg equivalent of Clinical Center Reference Endotoxin.
3. Have a body weight greater than 65 kg and a body mass index (BMI) below 30.
4. Have normal lung function, defined as:

   * Forced vital capacity (FVC) > 80% of that predicted value;
   * FEV1 > 80% of that predicted value; and
   * FEV1/FVC ratio > 80% of predicted values.
5. Have vital signs within the normal range, as follows:

   * Oral body temperature: 35.0 to 36.5 °C.
   * Blood pressure (BP):
   * After at least 3 minutes of rest, measured in the supine position:
   * Systolic BP: 90 to 140 mm Hg.
   * Diastolic BP: 50 to 90 mm Hg.
   * Then, after 1 minute standing:
   * Systolic BP: no more than a 20 mmHg decrease.
   * Diastolic BP: no more than a 10 mm Hg decrease.
   * Heart rate: after at least 3 minutes of rest and measured in the supine position: 40 to 90 beats per minute (bpm).
6. Have a hemoglobin level of 12.0 g/dL or more.
7. Have been a non-smoker for the preceding 12 months.
8. Willing and able to give written informed consent and to comply with the requirements of the study.
9. Female subjects must not be pregnant or lactating.
10. All subjects who are sexually active must use a medically acceptable and highly effective method of birth control for the duration of the study, and continue for 90 days after the end of treatment.

    -

Exclusion Criteria:

1. Have any condition, including findings in the medical history or in the pre-study assessments, which, in the opinion of the investigator, constitute a risk or contraindication for the participation of the subject to the study, or that could interfere with the study objectives, conduct, or evaluation including, but not limited to:

   * Any clinically significant abnormality in the results of pre-study safety laboratory tests.
   * A positive test for drugs of abuse or alcohol breath test.
   * Positive results from serum tests for Hepatitis B surface antigen (not due to vaccination), Hepatitis C, or Human Immunodeficiency Virus.
   * History or presence of lung disease including asthma, chronic obstructive lung disease, or emphysema.
   * History of atopy, including hay fever or atopic dermatitis.
   * History or presence of liver disease.
   * Hyperthyroidism, hypoglycemia, hyperglycemia, or diabetes mellitus.
   * History or presence of autoimmune disorders including myositis, hepatitis, idiopathic thrombocytopenic purpura, psoriasis, rheumatoid arthritis, interstitial nephritis, Sjögren's syndrome, thyroiditis, or systemic lupus erythaematosus.
   * Occurrence of any acute infection within the last 2 weeks before dosing.
2. Presence or history of any severe allergic reactions; or history of allergy to any medications that may be used or prescribed in the course of this study (eg, albuterol, prednisolone, acetaminophen, aspirin or other non-steroidal anti-inflammatory agents, or adalimumab).
3. History or presence of drug or alcohol abuse. (i;e. average daily intake of 3 units or a maximum weekly intake of greater than 21 units (1 unit equals 340 milliliters [ml] of beer, 115 ml of wine, or 43 ml of spirits).
4. History or active manifestation of a serious psychiatric illness including depression, suicidal ideation, or psychosis.
5. Positive test for latent tuberculosis.
6. Loss or donation of blood within 12 weeks prior to entry into the study, or plasma donation within 1 week prior to entry into the study.
7. Use of any prescription drugs within 2 weeks or over-the-counter medication, including herbal supplements or multivitamins, within 1 week before drug administration without prior approval from the investigator.
8. Use of any medication that may impact the results of any of the challenges, interfere with any other medications potentially used in the study, including steroids, beta blockers, or non-steroidal anti-inflammatory agents.
9. Previous participation in this study, or administration of any investigational drug within 12 weeks prior to entry into the study.
10. Exposure to endotoxin, within 12 weeks of signing the informed consent for this study.
11. History of exposure to keyhole limpet hemocyanin (KLH), dog rabies vaccine, or history of immunization with inactivated Hepatitis A virus.

    -

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
sputum cells count | 7 days

REFERENCES:
- [Derived] Michel O, Dinh PH, Doyen V, Corazza F. Anti-TNF inhibits the airways neutrophilic inflammation induced by inhaled endotoxin in human. BMC Pharmacol Toxicol. 2014 Nov 3;15:60. doi: 10.1186/2050-6511-15-60. PMID 25371053